CLINICAL TRIAL: NCT05758064
Title: How to Rescue Hormonal Replacement Frozen Embryo Transfer Cycle With Low Serum Progesterone? A Randomized Control Trial.
Brief Title: The Rescue of Hormonal Replacement Frozen Embryo Transfer Cycle With Low Serum Progesterone.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: El Shatby University Hospital for Obstetrics and Gynecology (Other)
Responsible Party: Principal Investigator, Aly Hussein, Principal investigator, El Shatby University Hospital for Obstetrics and Gynecology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0305825
Record Dates: First submitted 2023-02-08; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Hormonal Replacement Frozen Embryo Transfer Cycle
MeSH Terms: interventions — Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral dydrogesterone (Active Comparator): 60 patients in HRT frozen embryo transfer with low serum progesterone less than 10 ng/ml 24 hours before the embryo transfer will be given oral 10 mg dydrogesterone (Duphaston®, Abbott) twice daily
  Interventions: Drug: Duphaston
- subcutaneous progesterone (Active Comparator): 60 patients in HRT frozen embryo transfer with low serum progesterone less than 10 ng/ml 24 hours before the embryo transfer will be subcutaneous injection 25mg daily (Prolutex®, IBSA).
  Interventions: Drug: prolutex

INTERVENTIONS:
Drug: Duphaston — 10 mg tablet will be given twice
  Arms: Oral dydrogesterone
Drug: prolutex — subcutaneous injection daily
  Arms: subcutaneous progesterone

SUMMARY:
Frozen embryo transfer (FET) is increasingly adopted strategy in modern IVF. Among the many factors that have contributed to such change, the pursuit of an ovarian hyperstimulation syndrome free clinic has been strongly required. Improvements in the vitrification and warming processes and the excellent cryo-survival rates have turned FET in our main tool for preventing this complication. Moreover, a freeze all strategy has proven to provide excellent or even better pregnancy rates (PRs), not only in high but also in normal responders.

While ART have rapidly evolved in the areas of embryo culture, vitrification and understanding of the embryo development, little progress has been achieved regarding endometrial preparation for FET. Undoubtedly, correct implantation requires a good quality embryo and a suitable decidualized endometrium. Artificial cycles require hormone replacement treatment (HRT) with estradiol and progesterone (P4). However, there is not a single standardized treatment described for optimal endometrial preparation and no protocol has proven superiority in terms of reproductive outcomes.(5, 6) Although artificial preparation is the most convenient method to schedule FET cycles, recent reports have highlighted a potentially detrimental effect of low P4 levels prior to FET on miscarriage and live birth rates (LBRs). These results have been observed both in homologous and oocyte recipient FET cycles(7, 8), but also in FET cycles of embryos that had undergone PGT for aneuploidies (PGT-A).(9) Additional P4 supplementation may be a way to improve reproductive outcomes in these patients.

Our open labelled randomized control study aims to investigate whether patients with low serum P4 levels the day before FET under standard HRT can benefit in terms of clinical and ongoing pregnancy and implantation rates from an individualized luteal phase support consisting in the addition of oral dydrogesterone supplementation or daily subcutaneous P4 injection.

DETAILED DESCRIPTION:
A randomized control trial which will be conducted at El-Shatby University Maternity Hospital and private two private ART centres in Alexandria, Egypt.

120 patients in which HRT-FET cycles with low serum progesterone levels will divided into two groups :

* Group A: 60 patients will be given oral 10 mg dydrogesterone (Duphaston®, Abbott) twice daily or,
* Group B: 60 patients will be given subcutaneous injection 25mg daily (Prolutex®, IBSA).

METHODS Investigation Basal hormonal profile before initiation of treatment, a basal hormonal profile will be performed in all patients (basal FSH, LH, and estradiol levels) Pelvic ultrasound using a transvaginal probe, to assess ovaries, tubes and document uterine size, shape and endometrial thickness.

Endometrial preparation:

A transvaginal scan will be performed on the second day of the menstrual cycle to document baseline endometrial thickness.

HRT preparation of endometrium will be started day two of the cycle by administration of estradiol valerate at dose 8 mg daily.

The endometrial thickness and pattern will be assessed starting from day 10 of estradiol supplementation. If the endometrial thickness is less than 7 mm, oestradiol valerate administration will be continued and reassessed every 3 days up to 21days and if no improvement the cycle will be cancelled.

When the endometrial thickness reaches a minimum of 7 mm with a triple-line appearance, patients will start progesterone supplementation. Vaginal progesterone at a daily dose of 800 mg will administered (cyclogest suppository 400mg. twice daily). Blastocyst transfer will be done after 5 complete days of progesterone administration.

A morning serum progesterone level will be measured 24 hours before embryo transfer. If the serum progesterone level is bellow <10 ng/mL (1) rescue progesterone dose will be started before blastocyst transfer.

Patients with low serum progesterone will be randomized to receive extra progesterone supplementation in the form of either:

* Group A: oral 10 mg dydrogesterone (Duphaston®, Abbott) twice daily or,
* Group B: subcutaneous injection 25mg daily (Prolutex®, IBSA). The serum progesterone will be measured again on the day of embryo transfer and the day after.

The HRT will be continued until a pregnancy test is performed, and in cases of a positive pregnancy test, estradiol valerate and progesterone will be continued till week 10 of gestation.

III. Measuring the level of beta HCG:

The level of HCG will be measured for diagnosis of pregnancy 14 days after embryo transfer.

IV. Detection of Clinical pregnancy rate:

Transvaginal ultrasonography will be used to detect the appearance of the gestational sac with a fetal pole in the uterus two weeks after positive pregnancy test.

Cases will be followed up till the end of first trimester to detect abortion rate.

ELIGIBILITY:
Inclusion Criteria:

1. Patient prepared for frozen blastocyst transfer.
2. Maternal age ranges from less than 40 years.
3. BMI < 35kg/m2.
4. Normal uterine cavity.

Exclusion Criteria:

1. Uncorrected endometrial, uterine or pelvic pathology.
2. Recurrent implantation failure cases.
3. Patients suffering from recurrent miscarriages.
4. Male factor infertility due to azoospermia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | at the 6 th weeks of pregnancy
  percentage of cases in which observation of a gestational sac with fetal heart beat by transvaginal ultrasound at 6 weeks of pregnancy

SECONDARY OUTCOMES:
Serum progesterone level on the day of FET | on the day of embryo transfer(before transfer)
  Serum progesterone level on the day of FET
Implantation rate | at the 6 th week of pregnancy
  it is calculated as the number of intrauterine gestational sacs observed by transvaginal ultrasonography divided by the number of transferred embryos at the 6 th week of pregnancy and then multiplied by 100
Ongoing pregnancy rate | At the 20 th week of gestation
  Assessing the difference in the ongoing pregnancy rate when the pregnancy had completed ≥20 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Aly A Hussein, Dr, Study Chair — University of Alexandria
Locations (2):
- Egypt (2):
  - Elshatby University Maternity Hospital, Alexandria
  - Faculty of Medicine, University of Alexandria, Alexandria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Devroey P, Polyzos NP, Blockeel C. An OHSS-Free Clinic by segmentation of IVF treatment. Hum Reprod. 2011 Oct;26(10):2593-7. doi: 10.1093/humrep/der251. Epub 2011 Aug 9. PMID 21828116
- [Background] Chen ZJ, Shi Y, Sun Y, Zhang B, Liang X, Cao Y, Yang J, Liu J, Wei D, Weng N, Tian L, Hao C, Yang D, Zhou F, Shi J, Xu Y, Li J, Yan J, Qin Y, Zhao H, Zhang H, Legro RS. Fresh versus Frozen Embryos for Infertility in the Polycystic Ovary Syndrome. N Engl J Med. 2016 Aug 11;375(6):523-33. doi: 10.1056/NEJMoa1513873. PMID 27509101
- [Background] Wei D, Liu JY, Sun Y, Shi Y, Zhang B, Liu JQ, Tan J, Liang X, Cao Y, Wang Z, Qin Y, Zhao H, Zhou Y, Ren H, Hao G, Ling X, Zhao J, Zhang Y, Qi X, Zhang L, Deng X, Chen X, Zhu Y, Wang X, Tian LF, Lv Q, Ma X, Zhang H, Legro RS, Chen ZJ. Frozen versus fresh single blastocyst transfer in ovulatory women: a multicentre, randomised controlled trial. Lancet. 2019 Mar 30;393(10178):1310-1318. doi: 10.1016/S0140-6736(18)32843-5. Epub 2019 Feb 28. PMID 30827784
- [Background] Stormlund S, Sopa N, Zedeler A, Bogstad J, Praetorius L, Nielsen HS, Kitlinski ML, Skouby SO, Mikkelsen AL, Spangmose AL, Jeppesen JV, Khatibi A, la Cour Freiesleben N, Ziebe S, Polyzos NP, Bergh C, Humaidan P, Andersen AN, Lossl K, Pinborg A. Freeze-all versus fresh blastocyst transfer strategy during in vitro fertilisation in women with regular menstrual cycles: multicentre randomised controlled trial. BMJ. 2020 Aug 5;370:m2519. doi: 10.1136/bmj.m2519. PMID 32759285
- [Background] Ghobara T, Gelbaya TA, Ayeleke RO. Cycle regimens for frozen-thawed embryo transfer. Cochrane Database Syst Rev. 2017 Jul 5;7(7):CD003414. doi: 10.1002/14651858.CD003414.pub3. PMID 28675921
- [Background] Groenewoud ER, Cohlen BJ, Macklon NS. Programming the endometrium for deferred transfer of cryopreserved embryos: hormone replacement versus modified natural cycles. Fertil Steril. 2018 May;109(5):768-774. doi: 10.1016/j.fertnstert.2018.02.135. PMID 29778369
- [Background] Cedrin-Durnerin I, Isnard T, Mahdjoub S, Sonigo C, Seroka A, Comtet M, Herbemont C, Sifer C, Grynberg M. Serum progesterone concentration and live birth rate in frozen-thawed embryo transfers with hormonally prepared endometrium. Reprod Biomed Online. 2019 Mar;38(3):472-480. doi: 10.1016/j.rbmo.2018.11.026. Epub 2019 Jan 5. PMID 30642638
- [Background] Volovsky M, Pakes C, Rozen G, Polyakov A. Do serum progesterone levels on day of embryo transfer influence pregnancy outcomes in artificial frozen-thaw cycles? J Assist Reprod Genet. 2020 May;37(5):1129-1135. doi: 10.1007/s10815-020-01713-w. Epub 2020 Feb 10. PMID 32043182
- [Background] Gaggiotti-Marre S, Martinez F, Coll L, Garcia S, Alvarez M, Parriego M, Barri PN, Polyzos N, Coroleu B. Low serum progesterone the day prior to frozen embryo transfer of euploid embryos is associated with significant reduction in live birth rates. Gynecol Endocrinol. 2019 May;35(5):439-442. doi: 10.1080/09513590.2018.1534952. Epub 2018 Dec 26. PMID 30585507